CLINICAL TRIAL: NCT00319163
Title: An Open-label, Single-dose, Randomized, 2-period, Crossover, Bioequivalence Study to Compare Two Manufacturing Processes for Levonorgestrel 90 mg/Ethinyl Estradiol 20 mg (LNG/EE) in Healthy, Cycling Women
Brief Title: Study Comparing Two Manufacturing Processes for Levonorgestrel 90 mg/Ethinyl Estradiol 20 mg (LNG/EE) in Healthy, Cycling Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0858A2-108
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: oral contraceptive; therapeutic equivalency; contraceptives, oral, combined
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

INTERVENTIONS:
Drug: levonorgestrel/ethinyl estradiol

SUMMARY:
Primary Objective: To determine the bioequivalence between the clinical batch process and the new processes for manufacturing LNG/EE.

Secondary Objective: To obtain additional safety and tolerability data concerning LNG/EE in healthy, cycling women.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 - 35 years of age
* Non-smokers

Exclusion Criteria:

* History of thromboembolic disease
* Prior adverse experiences with oral contraceptives

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic sampling over the course of 4 days following two different formulations of the same compound

SECONDARY OUTCOMES:
Additional safety--clinical labs
electrocardiograms (ECGs)
vital signs
and adverse event recording over 4 days following administration of each formulation (LNG/EE)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Miami, Florida, United States